CLINICAL TRIAL: NCT05343182
Title: Vestibulectomy: A Prospective Comparison of Two Surgical Techniques for the Treatment of Provoked Localized Vulvodynia (PVD)
Brief Title: Vestibulectomy Surgical Techniques Comparison Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Catherine M Leclair, MD, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 24107
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vulvar Pain; Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Vestibulectomy (Active Comparator)
  Interventions: Other: Modified Technique
- Traditional Vestibulectomy (Active Comparator)
  Interventions: Other: Traditional Technique

INTERVENTIONS:
Other: Modified Technique — This operation is performed using modified anesthesia care/deep sedation (MAC) for anesthesia. The vestibule is removed to the boundary of Harts line. The surgical flap for this procedure is the Hymen plus 1 cm of the vagina.
  Arms: Modified Vestibulectomy
Other: Traditional Technique — This operation is performed using an Laryngeal Mask Airway (LAM), (modified anesthesia care/deep sedation) for anesthesia. The vestibule is removed 0.5 to 1 cm beyond the boundary of the Hart's line. The Hymen plus 1 cm of the vagina is excised.
  Arms: Traditional Vestibulectomy

SUMMARY:
Vestibulectomy Surgical Techniques Comparison Study

DETAILED DESCRIPTION:
Vestibulectomy: A Prospective Comparison of Two Surgical Techniques for the treatment of Provoked Localized Vulvodynia (PVD)

ELIGIBILITY:
Inclusion Criteria:

1. Reported provoked tenderness to the vestibule for at least 3 months in non-pregnant, estrogen-replete healthy subjects aged 18 years or over meeting Friedrich's criteria for PVD44-45 and supported by the ISSVD Terminology Consensus Definition45 for vulvar pain. Subjects who are >45years of age must have either have a maturation index52 of < 10% parabasal cells or willingness to participate in local estrogen replacement until achieving this same clinical result.
2. Cotton swab Test30-31 mean verbal rating score of ≥4/10 in 4 of 6 defined points of the vestibule (2, 4, 6, 8, 10, 12 o'clock) and cotton swab test verbal score ≤ 2/10 for the labia majora and minora, intra labial sulcus, and perineum
3. Ability to insert a regular Tampax® tampon
4. Baseline Tampon Test verbal pain score ≥430

f. Phone and internet access e. Willingness to engage in pelvic floor physical therapy (PT)

Exclusion Criteria:

1. Pregnancy
2. Any other clinical reason for dyspareunia (endometriosis pain, chronic pelvic pain, vulvar dermatoses such as psoriasis, lichen sclerosus)
3. Unable or unwilling to complete baseline assessments
4. Prior vestibulectomy or hymen surgery
5. Prior or current use of testosterone dosed for gender affirmation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Tampon Test pain scores from baseline to 3 months | Baseline visit to 3 months after surgery
  The change from baseline in pain measured by the Tampon Test at 3 months after surgery. The tampon test is a validated tool used to measure (vulva) vestibular skin pain by having participants insert and remove a tampon. Participants will be asked to rate their pain along a 100 mm Visual Analog Scale on a scale of 0 (No pain) to 10 (Pain as bad as you can imagine). This test will occur at baseline and 3 months follow up.
Change in pain scores from baseline to 6 months | Baseline visit to 6 months after surgery
  The change from baseline in pain measured by the Tampon Test at 6 months after surgery. The tampon test is a validated tool used to measure (vulva) vestibular skin pain by having participants insert and remove a tampon. Participants will be asked to rate their pain along a 100 mm Visual Analog Scale on a scale of 0 (No pain) to 10 (Pain as bad as you can imagine). This test will occur at baseline and 6 months follow up.
Change in pain scores from baseline to 12 months | Baseline visit to 12 months after surgery
  The change from baseline in pain measured by the Tampon Test at 12 months after surgery. The tampon test is a validated tool used to measure (vulva) vestibular skin pain by having participants insert and remove a tampon. Participants will be asked to rate their pain along a 100 mm Visual Analog Scale on a scale of 0 (No pain) to 10 (Pain as bad as you can imagine). This test will occur at baseline and 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Leclair, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States